CLINICAL TRIAL: NCT03107689
Title: Prospective Cohort Study of Intravenous Lipid Emulsion for Resuscitating Critically-ill Poisoned Patients
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: American College of Medical Toxicology (Other)
Responsible Party: Sponsor
Other Study IDs: HS-13-00634
Record Dates: First submitted 2016-01-12; First posted 2017-04-11 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-12

CONDITIONS: Overdose
Keywords: ILE; lipid; overdose; resuscitation
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: administration of intravenous lipid emulsion — all patients receive intravenous lipid emulsion at the discretion of the treating provider. This registry prospectively collects detailed information on such patients

SUMMARY:
The purpose of this project is to evaluate the case characteristics of patients who receive intravenous lipid emulsion therapy. Previous literature to date has focused on animal studies or has been primarily limited to case reports or small case series. This prospectively collected data set will permit a much more detailed description of the use of lipid, its potential benefits, and potential harms.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the case characteristics of patients who receive intravenous lipid emulsion therapy. A secondary objective is to determine the mortality in this critically ill population of individuals.

Previous literature to date has focused on animal studies or has been primarily limited to case reports or small case series. This prospectively collected data set will permit a much more detailed description of the use of lipid, its potential benefits, and potential harms.

ELIGIBILITY:
Inclusion Criteria:

* receiving intravenous lipid emulsion for treatment of a drug toxicity
* Evaluation of a medical toxicologist as part of the ToxIC registry consortium

Exclusion Criteria:

* not evaluated by a medical toxicologist participating in ToxIC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive intravenous lipid emulsion by a toxicologist, participating in the ToxIC registry, who complete the lipid subregistry
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Survival | Survival is measured at hospital discharge. The study is open to enrollment indefinitely. It is estimated approximately 100 subjects will be enrolled in 5 years
  The primary objective is to compare survival based on lipophilicity (as measured by LogD) of the drugs

CONTACTS AND LOCATIONS:
Overall Officials: michael levine, md, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - ACMT; ToxIC participating sites, Phoenix, Arizona
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No